CLINICAL TRIAL: NCT03853057
Title: The Effect of Positive Pressure and Body Position on Volumetric Capnography Assessed by Electrical Impedance Tomography
Brief Title: Positive Pressure and Gravity Affect Volumetric Capnography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 04112014
Record Dates: First submitted 2015-03-03; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2016-02

CONDITIONS: Hypoventilation
Keywords: volumetric capnography; gravity; mechanical ventilation; EIT
MeSH Terms: conditions — Hypoventilation | interventions — Posture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non-invasive ventilation (Experimental): Non-invasive positive pressure at different body positions: sitting - supine - prone - right lateral and left lateral.
  Interventions: Other: body positions

INTERVENTIONS:
Other: body positions — positive pressure ventilation at different body positions

SUMMARY:
Volumetric capnography is an interesting and non-invasive tool for monitoring ventilation in mechanically ventilated patients. The aim of this study was to test the effect of positive pressure ventilation and different body positions on volumetric capnograms.

DETAILED DESCRIPTION:
In this interventional study awake and healthy volunteers will be submitted to spontaneous, pressure support and control pressure ventilation using a tight nasal mask. Volumetric capnography and electrical impedance tomography (EIT) will be continuously recorded during the protocol. Different body positions were randomly tested. Analysis of global and regional distribution of ventilation using EIT will be matched with changes observed in volumetric capnography-derived parameters.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesia physical status I.
* Age between 25-39 years old,
* Body mass index between 23-28 kg/m2,
* Non-smokers.

Exclusion Criteria:

* Presence of pulmonary or cardiac diseases.
* Abnormal spirometry.

Ages: 28 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Analysis of the changes in volumetric capnographic parameters with changes in body positioning and positive pressure ventilation. | 4 hours
  The volunteers are breathing spontaneously with and without positive pressure support. Capnographic parameters were registered at each studied condition.

SECONDARY OUTCOMES:
Electrical impedance images of the distribution of ventilation with changes in body positioning and positive pressure ventilation. | 4 hours
  The volunteers are breathing spontaneously with and without positive pressure support. Electrical impedance images were taken at each studied condition.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo H Tusman, MD, Principal Investigator — Hospital Privado de Comunidad
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Tusman G, Scandurra A, Bohm SH, Suarez-Sipmann F, Clara F. Model fitting of volumetric capnograms improves calculations of airway dead space and slope of phase III. J Clin Monit Comput. 2009 Aug;23(4):197-206. doi: 10.1007/s10877-009-9182-z. Epub 2009 Jun 11. PMID 19517259